CLINICAL TRIAL: NCT03948958
Title: Pilot Trial to Assess Functional, Microbial, Radiological and Patient Reported Outcomes at Totally Implantable Venous Access Device (Port) Removal (PREMO Study)
Brief Title: PREMO Study: to Investigate Port REMoval Outcomes
Acronym: PREMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: B. Braun Medical SA (Industry)
Responsible Party: Principal Investigator, Stas Marguerite, Professor Doctor, Universitaire Ziekenhuizen KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: S62321
Record Dates: First submitted 2019-05-10; First posted 2019-05-14 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Neoplasms; Cystic Fibrosis
Keywords: Vascular Access Devices; Implantable port; Flush interval; Catheter function; Catheter-related infection; Catheter tip location; Catheter tip thrombus; Catheter sleeve; Patient-reported outcome measure
MeSH Terms: conditions — Neoplasms; Cystic Fibrosis; Catheter-Related Infections | interventions — Blood Coagulation; Patient Reported Outcome Measures; Catheters

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TIVAD evaluation (Experimental): TIVAD evaluation at port removal evaluation of catheter function, visualization of catheter tip, presence of thrombus material and sleeve and any device damage during linogram (contrast injection via TIVAD), tip and chamber content microbiological culture, macroscopic catheter and port chamber evaluation PROM: patient reported outcome measurements regarding TIVAD insertion, presence and removal
  Interventions: Other: Evaluation of the catheter function; Other: Catheter tip location, thrombus, sleeve and device damage visualization; Other: Catheter-related colonization; Other: patient-reported outcome measures (PROM) related to the presence of the TIVAD; Other: Macroscopic evaluation of the port chamber and catheter

INTERVENTIONS:
Other: Evaluation of the catheter function — Catheter function will be measured by the CINAS (Catheter injection and aspiration classification)
Other: Catheter tip location, thrombus, sleeve and device damage visualization — Catheter tip location, thrombus, sleeve and device damage will be visualized by linogram
Other: Catheter-related colonization — TIVAD colonization will be investigated by microbiological culture of the tip and chamber content
Other: patient-reported outcome measures (PROM) related to the presence of the TIVAD — PROM will evaluate patient's experiences regarding the TIVAD insertion, dwell time, and removal using the Leuven Patient Reported Experiences at Port removal (Leuven PREP) questionnaire.
Other: Macroscopic evaluation of the port chamber and catheter — Macroscopic evaluation of the port chamber and catheter will be performed after port removal.

SUMMARY:
A Totally Implantable Venous Access Device (TIVAD) that is no longer in use for intravenous therapy, should be flushed at established intervals to promote and maintain patency. No consensus has been established regarding the optimal duration of the interval between 2 maintenance sessions. This exploratory study will focus on catheter status under the current 3-monthly flush regimen.

DETAILED DESCRIPTION:
A Totally Implantable Venous Access Device (TIVAD) or so called implantable port that is no longer in use for intravenous therapy, should be removed or flushed at established intervals to promote and maintain patency. The maintenance procedure consists of a 10 ml 0.9% sodium chloride pulsatile flush. No consensus has been established regarding the optimal duration of the interval between 2 maintenance sessions. In het university hospitals Leuven the current interval is 3 months. Studies confirmed the safety and efficacy of an extended maintenance interval to once every 4 months. Many patients have relatively poor compliance with their regular port flushing procedure.

Clinicians tend to prolong the recommended interval or even to omit the maintenance procedure. Therefore in clinical practice, intervals vary widely among institutions. To the best of our knowledge, a comprehensive investigation of the risks related to catheter patency, bacterial colonization and catheter integrity, has never been performed in patients whose port is electively removed using a 3 months flushing maintenance regimen. To assess the impact of the maintenance interval, patients will be included in the study if the patient's TIVAD is not being used for regularly therapy for a total period of at least one year.

This exploratory study will focus on catheter function and colonisation, tip position and tip thrombosis, sleeve formation, removal problems and also patient experiences at elective planned TIVAD removal therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients of 18 years and older, with a TIVAD that is no longer used for intravenous therapy on a regular basis for the past 365 days after completing initially planned treatment.
* Patients planned for an elective TIVAD removal under local anaesthesia.
* Patients able to participate in the study and willing to sign an informed consent.
* Patients able to understand and read Dutch.

Exclusion Criteria:

• History of fever and/or chills following last flushing procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-07-08 (Actual)

PRIMARY OUTCOMES:
TIVAD function | during the 1 day of TIVAD removal, before the linogram
  will be assessed in terms of both injection and aspiration abilities. The ability is scored as easy, difficult or impossible along the Catheter Injection and Aspiration (CINAS) classification.

SECONDARY OUTCOMES:
Catheter tip position visualization by fluoroscopy | during the 1 day of TIVAD removal, just before the linogram
  The patient will be positioned in a nearly standing position with chest elevation of 17°
Port chamber filling, sleeve formation, sleeve extend, catheter tip thrombosis and damage in port chamber or catheter trajectory | during the 1 day of TIVAD removal
  will be visualised by linogram (digital substraction angiography)
Catheter tip and port chamber culture | during the 1 day of TIVAD removal (following TIVAD removal)
  microbial culture

OTHER OUTCOMES:
Patient-reported outcome measure | during the 1 day of TIVAD removal
  Patient's experiences will be collected by means of the Leuven Patient Reported Experiences at Port removal (Leuven PREP) questionnaire a self-reported 25-items questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Marguerite Stas, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goossens GA, Jerome M, Janssens C, Peetermans WE, Fieuws S, Moons P, Verschakelen J, Peerlinck K, Jacquemin M, Stas M. Comparing normal saline versus diluted heparin to lock non-valved totally implantable venous access devices in cancer patients: a randomised, non-inferiority, open trial. Ann Oncol. 2013 Jul;24(7):1892-1899. doi: 10.1093/annonc/mdt114. Epub 2013 Apr 3. PMID 23553060
- [Background] Odabas H, Ozdemir NY, Ziraman I, Aksoy S, Abali H, Oksuzoglu B, Isik M, Civelek B, Dede D, Zengin N. Effect of port-care frequency on venous port catheter-related complications in cancer patients. Int J Clin Oncol. 2014 Aug;19(4):761-6. doi: 10.1007/s10147-013-0609-7. Epub 2013 Aug 27. PMID 23978939
- [Background] Palese A, Baldassar D, Rupil A, Bonanni G, Capellari Maria T, Contessi D, De Crignis L, Vidoni A, Piller Roner S, Zanini A. Maintaining patency in totally implantable venous access devices (TIVAD): a time-to-event analysis of different lock irrigation intervals. Eur J Oncol Nurs. 2014 Feb;18(1):66-71. doi: 10.1016/j.ejon.2013.09.002. Epub 2013 Oct 4. PMID 24100090
- [Background] Diaz JA, Rai SN, Wu X, Chao JH, Dias AL, Kloecker GH. Phase II Trial on Extending the Maintenance Flushing Interval of Implanted Ports. J Oncol Pract. 2017 Jan;13(1):e22-e28. doi: 10.1200/JOP.2016.010843. Epub 2016 Oct 23. PMID 28084883
- [Background] Dal Molin A, Guerretta L, Mazzufero F, Rasero L. The management of totally implanted venous ports in the ambulatory oncologic patient. J Vasc Access. 2009 Jan-Mar;10(1):22-6. doi: 10.1177/112972980901000104. PMID 19340795
- [Background] Goossens GA. Flushing and Locking of Venous Catheters: Available Evidence and Evidence Deficit. Nurs Res Pract. 2015;2015:985686. doi: 10.1155/2015/985686. Epub 2015 May 14. PMID 26075094
- [Background] Ferroni A, Gaudin F, Guiffant G, Flaud P, Durussel JJ, Descamps P, Berche P, Nassif X, Merckx J. Pulsative flushing as a strategy to prevent bacterial colonization of vascular access devices. Med Devices (Auckl). 2014 Nov 7;7:379-83. doi: 10.2147/MDER.S71217. eCollection 2014. PMID 25404862
- [Background] Gristina AG, Giridhar G, Gabriel BL, Naylor PT, Myrvik QN. Cell biology and molecular mechanisms in artificial device infections. Int J Artif Organs. 1993 Nov;16(11):755-63. PMID 8150521
- [Background] Douard MC, Arlet G, Longuet P, Troje C, Rouveau M, Ponscarme D, Eurin B. Diagnosis of venous access port-related infections. Clin Infect Dis. 1999 Nov;29(5):1197-202. doi: 10.1086/313444. PMID 10524963
- [Background] Brouns F, Schuermans A, Verhaegen J, De Wever I, Stas M. Infection assessment of totally implanted long-term venous access devices. J Vasc Access. 2006 Jan-Mar;7(1):24-8. doi: 10.1177/112972980600700105. PMID 16596525
- [Background] Tang S, Beigel R, Arsanjani R, Larson B, Luthringer D, Siegel R. Infective Endovascular Fibrin Sheath Vegetations-A New Cause of Bacteremia Detected by Transesophageal Echocardiogram. Am J Med. 2015 Sep;128(9):1029-38. doi: 10.1016/j.amjmed.2015.03.019. Epub 2015 Apr 10. PMID 25865922
- [Background] Onal B, Coskun B, Karabulut R, Ilgit ET, Turkyilmaz Z, Sonmez K. Interventional radiological retrieval of embolized vascular access device fragments. Diagn Interv Radiol. 2012 Jan-Feb;18(1):87-91. doi: 10.4261/1305-3825.DIR.4098-10.1. Epub 2011 Feb 8. PMID 21305467
- [Background] Kojima S, Hiraki T, Gobara H, Iguchi T, Fujiwara H, Matsui Y, Mitsuhashi T, Kanazawa S. Fracture of totally implanted central venous access devices: a propensity-score-matched comparison of risks for Groshong silicone versus polyurethane catheters. J Vasc Access. 2016 Nov 2;17(6):535-541. doi: 10.5301/jva.5000606. Epub 2016 Oct 21. PMID 27768210
- [Background] Goossens GA, De Waele Y, Jerome M, Fieuws S, Janssens C, Stas M, Moons P. Diagnostic accuracy of the Catheter Injection and Aspiration (CINAS) classification for assessing the function of totally implantable venous access devices. Support Care Cancer. 2016 Feb;24(2):755-761. doi: 10.1007/s00520-015-2839-x. Epub 2015 Jul 26. PMID 26209949
- [Background] Bouza E, Martin-Rabadan P, Echenagusia A, Camunez F, Rodriguez-Rosales G, Simo G, Echenagusia M, Guembe M; GEIDI study group. Diagnosis of venous access port colonization requires cultures from multiple sites: should guidelines be amended? Diagn Microbiol Infect Dis. 2014 Feb;78(2):162-7. doi: 10.1016/j.diagmicrobio.2013.11.004. Epub 2013 Nov 14. PMID 24316016
- [Background] Marcy PY, Dahlet C, Brenet O, Yazbec G, Dubois PY, Salm B, Fouche Y, Mari V, Montastruc M, Lebrec N, Ancel B, Paillocher N, Dupoiron D, Rangeard O, Michel C, Chateau Y, Ettaiche M, Ferrero JM, Chamorey E. [Multicenter validation study of a questionnaire assessing patient satisfaction with and acceptance of totally-implanted central venous access devices]. Bull Cancer. 2015 Apr;102(4):301-15. doi: 10.1016/j.bulcan.2015.02.012. Epub 2015 Mar 21. French. PMID 25799876
- [Background] Goossens GA, Vrebos M, De Wever I, Stas M. Vacutainer filling time through subcutaneous venous access devices. J Vasc Access. 2004 Oct-Dec;5(4):154-60. doi: 10.1177/112972980400500404. PMID 16596559
- [Derived] Goossens GA, Douchy T, Jerome M, Peeters Y, Hompes D, Boecxstaens V. Port REMoval Outcomes (PREMO) study: Patients' experiences with a Totally Implantable Venous Access Device: A questionnaire at device removal. J Vasc Access. 2025 May 27:11297298251340461. doi: 10.1177/11297298251340461. Online ahead of print. PMID 40421915
- [Derived] Douchy T, Hompes D, Maleux G, Jerome M, Peeters Y, Goossens GA, Boecxstaens V. Port REMoval Outcomes (PREMO) study: A pilot study for functional, microbial, radiological, and macroscopic assessment of totally implantable venous access devices. J Vasc Access. 2025 May 13:11297298251335416. doi: 10.1177/11297298251335416. Online ahead of print. PMID 40359084